CLINICAL TRIAL: NCT06369064
Title: Comparison of the Effectiveness of Continuous Veno-venous Hemodialysis and Continuous Veno-venous Hemodiafiltration on Urea Reduction Rate in Intensive Care Patients With Acute Renal Injury : a Monocentric Controled Randomized Non Inferiority Open Labeled Study
Brief Title: Continuous Veno-venous Hemodialysis and Continuous Veno-venous Hemodiafiltration on Urea Reduction Rate in Intensive Care Patient
Acronym: CompEER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023A02707-38
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Acute Kidney Injury; Continuous Renal Replacement Therapy; Intensive Care Unit
Keywords: continuous venovenous hemodiafiltration; continuous venovenous hemodialysis; urea reduction rate
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CVVHD (Experimental): Patient requiring renal remplacement therapy treated with by continuous venovenous hemodialysis (CVVHD) method.
  Interventions: Other: CVVHD Dialysis parameters
- CVVHDF (Active Comparator): Patient requiring renal remplacement therapy treated with by continuous venovenous hemodiafiltration (CVVHDF) method.
  Interventions: Other: CVVHDF Dialysis parameters

INTERVENTIONS:
Other: CVVHD Dialysis parameters — Patients will receive a CVVHD dialysis with a dose of 25ml/kg/h dialysate (100% dialysate), with Fresenius Medical Care multiFiltrate PRO kit and Ultraflux AV1000S filter (polysuflone 1.8m²).Regional anticoagulation with citrate
  Arms: CVVHD
Other: CVVHDF Dialysis parameters — Patients will receive a CVVHDF dialysis with a dose of 25ml/kg/h dialysate (50% ultrafiltration, 50% dialysate), with Fresenius Medical Care multiFiltrate PRO kit and Ultraflux AV1000S filter (polysuflone 1.8m²). Systemic anticoagulation with heparine
  Arms: CVVHDF

SUMMARY:
In patients requiring renal replacement therapy (RRT) in the intensive care unit (ICU), continuous techniques are predominantly using due to better hemodynamic tolerance. The most employed techniques in ICU are continuous venovenous hemodiafiltration (CVVHDF) and continuous venovenous hemodialysis (CVVHD).

To our knowledge, there are no prospective studies comparing the efficiency of these two techniques with the same dose of dialysis (and the same filter).

In the CompEER study, we aim to compare the efficiency of CVVHD and CVVHDF on urea reduction rate in intensive care patients with acute kidney injury.

The research hypothesis is that CVVHD citrate technique is as effective as CVVHDF heparin technique for urea reduction and provides prolonged and stable clearance, facilitating antibiotic management during RRT.

DETAILED DESCRIPTION:
Acute Kidney Injury (AKI) is found in more than 50% of intensive care unit (ICU) patients, with 30% classified as AKI Network (AKIN) stage 3. Approximately 23% of AKI patients undergo RRT, predominantly utilizing continuous techniques due to better hemodynamic tolerance in unstable patients. Common continuous RRT techniques include continuous venovenous hemofiltration (CVVH), continuous venovenous hemodialysis (CVVHD), and continuous venovenous hemodiafiltration (CVVHDF).

The two most employed techniques in ICU are CVVHDF and CVVHD. However, the choice often depends on institutional practices rather than scientific evidence. Limited studies comparing these techniques at equivalent doses exist, and French recommendations allow intensivists discretion based on availability and team experience. A small, randomized study comparing different exchange rates found higher urea reduction in CVVHDF but lacked statistical significance. Current practices in ICU involve using CVVHDF with systemic anticoagulation or CVVHD with regional citrate anticoagulation based on practitioner preferences.

Despite potential benefits of CVVHD with citrate, such as extended filter lifespan and stable dialysis dose, the impact on concomitant treatments, especially antibiotics, needs consideration.

The study aims to demonstrate the non-inferiority of citrate-based continuous hemodialysis (CVVHD) compared to heparin-based continuous hemodiafiltration (CVVHDF) in terms of urea reduction rate at 24 hours in AKI patients requiring renal replacement therapy.

The hypothesis is that CVVHD citrate is as effective as CVVHDF heparin, providing prolonged and stable clearance, facilitating antibiotic management during RRT.

ELIGIBILITY:
Inclusion criteria:

* Adult patients hospitalized in ICU
* Undergo RRT session because of AKI stage 3
* At least one among criteria: pH < 7,20 / Blood urea > 30mM / Fluid overload uncontrolled by diuretics.
* Patient having given free and informed consent, and having signed the consent form or patient included in an emergency situation
* Patient affiliated with Social Security.

Exclusion criteria:

* End-stage chronic kidney disease on dialysis
* Intoxication with a dialyzable toxin (lithium
* Criteria for emergency dialysis initiation: hyperkaliemia >6,5mM with electrocardiographic signs
* Medical contraindication to regional citrate: severe liver failure
* Medical contraindication to anticoagulation or heparin anticoagulation: heparin induced thrombopenia or uncontrolled bleeding
* Pregnant women, parturient or breast-feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
urea reduction rate (URR) | 24 hours
  The primary endpoint is the rate of urea reduction (TRU) at 24h as a percentage TRU H24 = (urea rate at H0 - urea rate at H24) / urea rate at H0 in each arm.

SECONDARY OUTCOMES:
Creatinine clearance at H24 | 24 hours
  Measured Creatinine clearance at 24 hours (ml/min)
Urea clearance at H24 | 24 hours
  Measured Urea clearance at 24 hours (ml/min)
Urea clearance at H48 | 48 hours
  Measured Urea clearance at 48 hours (ml/min)
ICU Mortality | End of ICU Stay
  Number of patients who died while in ICU
Mortality at Day 28 | Day 28
  Number of patients who died betwwen day à and day 28
Organ failure-free days at Day 28 | Day 28
  Number of organ failure-free days at Day 28
Hypokalemia at Day 28 | Day 28
  Hypokalemia < 3mmol/l occurring between Day 0 and Day 28
Hypophosphatemia at Day 28 | Day 28
  Hypophosphatemia < 0.8mmol/l occurring between Day 0 and Day 28
Hypomagnesemia at Day 28 | Day 28
  Hypomagnesemia < 0.8mmol/l occurring between Day 0 and Day 28
Hyperkalemia at Day 28 | Day 28
  Hyperkalemia >6mmol/l occurring between Day 0 and Day 28
Medical Cost | 24 hours
  Cost of one continuous hemodialysis (CVVHD) session with citrate compared to one continuous hemodiafiltration (CVVHDF)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Roger, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

REFERENCES:
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Joannes-Boyau O, Honore PM, Perez P, Bagshaw SM, Grand H, Canivet JL, Dewitte A, Flamens C, Pujol W, Grandoulier AS, Fleureau C, Jacobs R, Broux C, Floch H, Branchard O, Franck S, Roze H, Collin V, Boer W, Calderon J, Gauche B, Spapen HD, Janvier G, Ouattara A. High-volume versus standard-volume haemofiltration for septic shock patients with acute kidney injury (IVOIRE study): a multicentre randomized controlled trial. Intensive Care Med. 2013 Sep;39(9):1535-46. doi: 10.1007/s00134-013-2967-z. Epub 2013 Jun 6. PMID 23740278
- [Background] Vinsonneau C, Allain-Launay E, Blayau C, Darmon M, Ducheyron D, Gaillot T, Honore PM, Javouhey E, Krummel T, Lahoche A, Letacon S, Legrand M, Monchi M, Ridel C, Robert R, Schortgen F, Souweine B, Vaillant P, Velly L, Osman D, Van Vong L. Renal replacement therapy in adult and pediatric intensive care : Recommendations by an expert panel from the French Intensive Care Society (SRLF) with the French Society of Anesthesia Intensive Care (SFAR) French Group for Pediatric Intensive Care Emergencies (GFRUP) the French Dialysis Society (SFD). Ann Intensive Care. 2015 Dec;5(1):58. doi: 10.1186/s13613-015-0093-5. Epub 2015 Dec 30. PMID 26714808
- [Background] Guilhaumou R, Benaboud S, Bennis Y, Dahyot-Fizelier C, Dailly E, Gandia P, Goutelle S, Lefeuvre S, Mongardon N, Roger C, Scala-Bertola J, Lemaitre F, Garnier M. Optimization of the treatment with beta-lactam antibiotics in critically ill patients-guidelines from the French Society of Pharmacology and Therapeutics (Societe Francaise de Pharmacologie et Therapeutique-SFPT) and the French Society of Anaesthesia and Intensive Care Medicine (Societe Francaise d'Anesthesie et Reanimation-SFAR). Crit Care. 2019 Mar 29;23(1):104. doi: 10.1186/s13054-019-2378-9. PMID 30925922
- [Background] Zarbock A, Kullmar M, Kindgen-Milles D, Wempe C, Gerss J, Brandenburger T, Dimski T, Tyczynski B, Jahn M, Mulling N, Mehrlander M, Rosenberger P, Marx G, Simon TP, Jaschinski U, Deetjen P, Putensen C, Schewe JC, Kluge S, Jarczak D, Slowinski T, Bodenstein M, Meybohm P, Wirtz S, Moerer O, Kortgen A, Simon P, Bagshaw SM, Kellum JA, Meersch M; RICH Investigators and the Sepnet Trial Group. Effect of Regional Citrate Anticoagulation vs Systemic Heparin Anticoagulation During Continuous Kidney Replacement Therapy on Dialysis Filter Life Span and Mortality Among Critically Ill Patients With Acute Kidney Injury: A Randomized Clinical Trial. JAMA. 2020 Oct 27;324(16):1629-1639. doi: 10.1001/jama.2020.18618. PMID 33095849